CLINICAL TRIAL: NCT04751643
Title: Assessment of Therapeutic Plasma Exchange to Improve Respiratory Function by Alleviating Cytokine Storm During Severe Covid-19 Infections Randomised Open-label Controlled Trial
Brief Title: Therapeutic Plasma Exchange to Alleviate Hyperinflammatory Condition During Severe Covid-19 Infections
Acronym: CovidEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0518; 2020-A03039-30 (Other: ID-RCB)
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care Units; ARDS, Human; Covid19
Keywords: Covid19; Therapeutic plasma exchange; Cytokine storm; Hyperinflammatory condition; Anti-IFN antibodies
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPE + usual treatments in intensive care unit according to the current state of knowledge. (Experimental): TPE + usual treatments in intensive care unit according to the current state of knowledge : 3 TPE sessions i.e. one per day during 3 consecutive days on day 1-3 (day 0 = inclusion Visit date)) + usual treatments in intensive care unit.
  Usual treatments of patients in intensive care unit with hyperinflammatory condition due to Covid-19 infection consist in supporting respiratory function, oxygen supplementation, non invasive ventilation, invasive ventilation, antibiotic, vasopressive support and corticosteroids (in absence of bacterial secondary infection)
  Interventions: Other: Therapeutic plasma exchange : 3 sessions in 3 consecutive days (day 1 to day 3); Other: Usual treatments in intensive care unit according to the current state of knowledge
- Usual treatments in intensive care unit according to the current state of knowledge (Active Comparator): Usual treatments of patients in intensive care unit with hyperinflammatory condition due to Covid-19 infection consist in supporting respiratory function, oxygen supplementation, non invasive ventilation, invasive ventilation, antibiotic, vasopressive support and corticosteroids (in absence of bacterial secondary infection)
  Interventions: Other: Usual treatments in intensive care unit according to the current state of knowledge

INTERVENTIONS:
Other: Therapeutic plasma exchange : 3 sessions in 3 consecutive days (day 1 to day 3) — Therapeutic plasma exchange (TPE) ; 3 sessions in 3 consecutive days (Day 1 to Day 3) in intensive care unit in addition to usual treatments.
  Plasma removed is replaced by thawed fresh frozen plasma. Plasma blood volume exchanged : 1.2 Apheresis type: centrifugation
  Arms: TPE + usual treatments in intensive care unit according to the current state of knowledge.
Other: Usual treatments in intensive care unit according to the current state of knowledge — Usual treatments of patients in intensive care unit with hyperinflammatory condition due to Covid-19 infection consist in supporting respiratory function, oxygen supplementation, non invasive ventilation, invasive ventilation, antibiotic, vasopressive support and corticosteroids (in absence of bacterial secondary infection)

SUMMARY:
Severe Covid-19 (Coronavirus Disease 2019) infections generate major but inappropriate production of cytokines and, in some cases, generate anti-IFN (Interferon) auto-antibodies, inducing acute respiratory distress syndrom (ARDS). Therapeutic plasma exchange (TPE) have been reported to be efficient for improving the hyperinflammatory condition state and the respiratory function, which has been described in case reports or small series.

The study aims to remove cytokines during cytokine storm and anti-IFN auto-antibodies (when present) to prevent developpement of an inappropriate immune response and to improve the clinical response to reanimation treatment, in particular the respiratory parameters leading to a rapid improvement of clinical status. To that aim, the study investigates to compare a treatment using TPE plus usual treatments in intensive care unit (experimental arm) versus usual treatments in intensive care unit (routine arm) in a randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized for COVID-19 confirmed by Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) or scanner
* Patients with PaO2/FiO2 between 75 and 175 mmHg requiring non invasive ventilation or high flow oxygen
* peripheral venous state allowing PE to be performed, according to the investigator's judgement, or possibility of placing a Sheldon-type veinous central line
* At least two biological results suggesting a cytokine storm or hyperinflammatory condition state among : C-reactive protéine (CRP)>50mg/L, Procalcitonin (PCT)>1µg/L, Fibrinogen>5g/L, D-dimer >1000ng/mL, Ferritin > 800ng/mL during the last 72 hours.
* Treatment with corticosteroids (at least 2 intakes of dexamethasone 6 mg or equivalent with another form of corticosteroids)
* Patient affiliated to a social security or similar scheme
* Information and written consent from the patient or if not possible from a confident person

Exclusion Criteria:

* Ventilated intubated patients
* Patient with advanced cancer and without curative possibility
* Bacterial or viral (HIV) infection explaining the worsening (the main reason)
* Body Mass Index > 40
* Severe hemodynamic instability with mean arterial pressure < 65 mmHg (whatever the noradrenaline dosage used)
* Known Immunoglobulin A (IgA) deficiency with anti-IgA antibodies
* Inclusion in another study that could interact with the Covidep study (investigator's judgement)
* Patient under legal protection measure
* Pregnant or breastfeeding women
* In case of allergy to amotosalen (psoralens) or AI-FFP (Amotosalen Inactivated Fresh Frozen Plasma) , use Se-FFP (Secured Fresh Frozen Plasma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Use of intubation and invasive ventilation (IV) between Day 0 (Inclusion Visit) and Day 10 | At day 10
  Proportion of patients requiring intubation between Day 0 and Day 10. Intubation use will be measured in both arms at Day 10.

SECONDARY OUTCOMES:
Assess the adverse events according to CTCAE v5.0 | Throughout the study : Day 1 to Day 10 and to the end of the study (Day 60 +/- 2 days)
  Adverse events according to CTCAE v5.0 measured throughout the study, in both groups, including tolerance to TPEs in the experimental group over the course of the study sessions.
PaO2/FIO2 (Partial Pressure of Oxygen/Fraction of Inspired Oxygen) (mmHg) at day 4 after inclusion (PaO2/FiO2 is a usual parameter for assessing evolution of ARDS) | At Day 4
  PaO2/FIO2 (mmHg) at day 4 after inclusion. This parameter will be compared between day 4 and day 0.The change corresponds to an increase of PaO2/FIO2 ratio equal or superior than 20%. The proportion of patients with a PaO2/FiO2 change at Day 4 will be compared between both arms.
Percentage of patients weaned from non invasive ventilation | At day 10
  Percentage of patients weaned from high flow oxygen. This parameter is compared between both arms (experimental and control arms).
O2 weaning capacity and duration of O2 dependence | At day 60
  This parameter is compared between both arms (experimental and control arms).
Survival at day 10 | At day 10
  Percentage of patients alive at day 10 after inclusion. This parameter is compared between both arms.
Survival at 2 months | At day 60 (+/- 2 days)
  Percentage of patients alive at 2 months after inclusion. This parameter is compared between both arms.
Percentage of patients without any increase in inflammatory parameters (analysis of C-reactive protein, Fibrinogen,D-Dimers, procalcitonin, Ferritin) | At day 4
  Percentage of patients without any increase in inflammatory parameters (analysis of C-reactive protein, Fibrinogen,D-Dimers, procalcitonin, Ferritin ) at day 4 compared to values at day 0. This parameter is compared between both arms.
Variation in cytokine and chemokine levels in the cytokine storm | At day 4
  Percentage of patients without any increase in cytokine or chemokine levels. Leucocyte and platelet cytokine or chemokine levels in ng/ml are assessed in both arms. Analysis of the entire panel of cytokines or chemokines defines an improvement or not. Comparison between both arms.
Percentage of patients with improved phenotype (decreased phenotype of exhausted cells) and improved function (improved proliferation) | At day 7
  Lymphocyte and NK (Natural Killer) labeling and analysis by flow cytometry at day 0 and day 7. Analysis of lymphocyte proliferation (after stimulation) at day 0 and day 7. Analysis of percentage of patients with improved phenotype (decreased phenotype of exhausted cells) and improved function (improved proliferation) ; this parameter is compared between both arms.
Percentage of patients with decreased platelet activation | At Day 4
  Phenotype of platelets and flow cytometry analysis performed before and after TPE or usual treatment. Percentage of patients with decreased platelet activation at day 4 ; this parameter is compared between both arms.
Percentage of patients with decreased platelet activation | At Day 7
  Phenotype of platelets and flow cytometry analysis performed before and after TPE or usual treatment. Percentage of patients with decreased platelet activation at day 7 ; this parameter is compared between both arms.
Change in anti-IFN auto-antibodies type I (α and ω) level | Day 0 and Day 4
  Change in anti-IFN auto-antibodies type I (α and ω) level at day 0 and day 4.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HEQUET, MD, PhD, Principal Investigator — Hospices Civils de Lyon - Etablissement Français du Sang
Locations (8):
- France (8):
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Croix Rousse, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Groupement Hospitalier Porte de Valence - Montélimar, Montélimar
  - Hôpital Pitié Salpétrière - Assistante Publique des Hôpitaux de Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Medipole Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guironnet-Paquet A, Hamzeh-Cognasse H, Berard F, Cognasse F, Richard JC, Yonis H, Mezidi M, Desebbe O, Delannoy B, Demeret S, Marois C, Saheb S, Le QV, Schoeffler M, Pugliesi PS, Debord S, Bastard P, Cobat A, Casanova JL, Pescarmona R, Viel S, Nicolas JF, Nosbaum A, Vocanson M, Hequet O. Therapeutic plasma exchange accelerates immune cell recovery in severe COVID-19. Front Immunol. 2025 Jan 17;15:1492672. doi: 10.3389/fimmu.2024.1492672. eCollection 2024. PMID 39896810